CLINICAL TRIAL: NCT01341951
Title: G-CSF in Acute Liver Failure and Alcoholic Hepatitis - A Pilot Study
Brief Title: Granulocyte Colony Stimulating Factor (G-CSF) in Acute Liver Failure and Alcoholic Hepatitis
Acronym: G-CSF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Dr. Virendra Singh, Postgraduate Institute of Medical Education and Research, Chandigarh, India
Organization: PIMERIndia (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIMERIndia
Record Dates: First submitted 2011-04-15; First posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-01

CONDITIONS: Liver Failure, Acute
Keywords: liver failure, Acute
MeSH Terms: conditions — Liver Failure, Acute | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-CSF therapy in acute liver failure and alcoholic hepatitis (Experimental): G-CSF therapy given in cases with acute liver failure and alcoholic hepatitis
  Interventions: Drug: Granulocyte colony stimulating factor

INTERVENTIONS:
Drug: Granulocyte colony stimulating factor — 300 I.U twice daily for 5 days

SUMMARY:
Granulocyte colony stimulating factor in acute liver failure and alcoholic hepatitis

DETAILED DESCRIPTION:
In this study 4 groups have been taken. Two groups of cases including Alcoholic patients and acute liver failure which are given G-CSF therapy and two groups of controls given standard therapy. Primary end point is to see the mobilization of CD-34 hematopoietic cells and survival. Secondary end point is to see the clinical and biochemical improvement in liver functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Liver failure as defined by AASLD.65
* Patients with Alcoholic hepatitis defined as follows: decades of heavy alcohol use (mean intake, approximately 100 g per day).The combination of an aspartate aminotransferase level that is elevated (but <300 IU per milliliter) and a ratio of the aspartate aminotransferase level to the alanine aminotransferase level that is more than 2, a total serum bilirubin level of more than 5 mg per deciliter (86 μmol per liter), an elevated INR, and neutrophilia.

Exclusion Criteria:

• Known hypersensitivity to filgrastim

* creatinine > 150 µmol/L
* infection or hemorrhage within the last 10 days
* documented hepatocellular carcinoma
* hepatitis B,C or human immunodeficiency virus seropositivity and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
• Mobilization of CD34 cells in the peripheral blood, a surrogate marker for hematopoietic stem cell mobilization | 1 year

SECONDARY OUTCOMES:
clinical and biochemical improvement in liver functions | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: virendra singh, Principal Investigator — Postgraduate Institute of Medical Education and Research Chandigarh India
Locations (1):
- Postgraduate Institute of Medical Education & Research Chandigarh India, Chandigarh, Chandigarh, India

REFERENCES:
- [Background] Spahr L, Lambert JF, Rubbia-Brandt L, Chalandon Y, Frossard JL, Giostra E, Hadengue A. Granulocyte-colony stimulating factor induces proliferation of hepatic progenitors in alcoholic steatohepatitis: a randomized trial. Hepatology. 2008 Jul;48(1):221-9. doi: 10.1002/hep.22317. PMID 18537187